CLINICAL TRIAL: NCT01666795
Title: Autoantibody Specificity and Response to Intravenous Immunoglobulin G (IVIG) in Immune Thrombocytopenia (ITP): a Retrospective Cohort Study
Brief Title: Autoantibody Specificity and Response to IVIG in ITP
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Second Affiliated Hospital of Medical College Shandong University (Other); Jinan Military General Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Ming Hou, Director, Department of Hematology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: ITP-006
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2012-08

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IVIG therapy in ITP: IVIG therapy in untreated adults with severe ITP

SUMMARY:
The objective of this human study was to evaluate the association between the specificity of anti-platelet autoantibodies and response to IVIG treatment.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a common autoimmune bleeding disorder, in which platelet surface GPIIb/IIIa and GPIb/IX are the two most frequently targeted autoantigens. Our previous studies in animal models of ITP demonstrated that intravenous immunoglobulin G (IVIG) could protect against anti-GPIIb/IIIa-mediated thrombocytopenia but failed to ameliorate ITP induced by most anti-GPIb/IX antibodies. The objective of this human study was to evaluate the association between the specificity of anti-platelet autoantibodies and response to IVIG treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) the diagnosis of ITP was based on the presence of isolated thrombocytopenia and the absence of any obvious initiating and/or underlying cause of the thrombocytopenia in accordance with the recently released international consensus guidelines,(2) a diagnosis was established during the 4 weeks prior to initiation of IVIG treatment, (3) age ≥ 18 years, (4) a platelet count of ≤ 20 × 109/L, and (5) a bleeding score ≥ 9 at the time of admission according to the clinical scoring system described by Khellaf et al. to assess the severity of hemorrhage.

Exclusion Criteria:

* a history of any ITP-specific treatment administered prior to or concomitantly with the IVIG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with severe ITP who underwent IVIG therapy and had platelet autoantibodies assayed
Sampling Method: Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2005-02; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
initial response | within 7 days of dosing
  The criteria for an initial response was a platelet count ≥ 30 × 109/L and doubling of the baseline count within 7 days of dosing (confirmed on at least 2 separate occasions at least 7 days apart), and absence of bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng J, Ma SH, Liu J, Hou Y, Liu XM, Niu T, Xu RR, Guo CS, Wang XM, Cheng YF, Ni H, Hou M. Association of autoantibody specificity and response to intravenous immunoglobulin G therapy in immune thrombocytopenia: a multicenter cohort study. J Thromb Haemost. 2014 Apr;12(4):497-504. doi: 10.1111/jth.12524. PMID 24517219